CLINICAL TRIAL: NCT05756868
Title: The Effect of Time-Restricted Feeding Intervention on Anthropometric Measurements, Biochemical Parameters, Diet Quality and Eating Behavior in Overweight Female Individuals
Brief Title: The Effect of Time-Restricted Feeding on Anthropometry, Biochemical Parameters, Diet Quality and Eating Behavior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Ayşen Yıldırım, Dietitian (MSc), Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AYildirim
Record Dates: First submitted 2022-11-25; First posted 2023-03-06 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-02

CONDITIONS: Fasting
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time restricted feeding (Experimental): The participants in the intervention group will receive a time restricted feeding intervention (first meal at 10:00, last meal at 18:00) for 6 weeks. Meals of the participants are planned as 8 hours of eating and 16 hours of fasting.
  Interventions: Behavioral: Time restricted feeding
- Control (No Intervention): Participants in the control group will not receive any dietary intervention. All participants were asked to continue in the same way they were fed before starting the study throughout the study.

INTERVENTIONS:
Behavioral: Time restricted feeding — In the time-restricted nutrition intervention, the first meal is scheduled at 10:00 and the last meal at 18:00 (ad libitum). Eating for 8 hours and fasting for 16 hours are targeted.
  Arms: Time restricted feeding

SUMMARY:
The goal of this randomized controlled trial is to to determine the effects of time-restricted feeding intervention on body weight, body composition, biochemical parameters and eating behaviors in overweight female individuals.

The main questions it aims to answer are:

1. Does time-restricted feeding intervention reduce daily energy intake?
2. Does time-restricted dietary intervention result in body weight and body fat loss?
3. Does time-limited nutritional intervention lead to improvements in biochemical parameters?
4. Does time-restricted feeding intervention improve eating behavior and eating awareness?
5. Does time-restricted feeding intervention adversely affect diet quality?

The participants in the intervention group will receive a time restricted feeding intervention (first meal at 10:00, last meal at 18:00) for 6 weeks. Meals of the participants are planned as 8 hours of eating and 16 hours of fasting.

Participants in the control group will not receive any dietary intervention.

DETAILED DESCRIPTION:
Following the ethics committee approval, the study will be carried out with the participants who applied to the Famagusta State Hospital Internal Medicine Polyclinic, Specialist Umut Hakligil.

In order to start the study, TR Ministry of Health Nicosia Dr. Necessary permissions were obtained from the Ethics Committee of Burhan Nalbantoğlu State Hospital.

The study is planned to be conducted with 40 female participants, who were not diagnosed with any disease by the physician, aged 19-65, slightly obese, with a BMI of 24.9-29.9 kg/m².

Before being included in the research, participants will be informed about the purpose of the research and the applications to be made during the research.

This information was supported with the valid consent form.

Data Collection Tool: A questionnaire form developed in line with the research purpose was used as a data collection tool in the research.

While collecting data on the individuals participating in the research, the "face-to-face interview method" (mask and distance due to the covid-19 pandemic) by taking necessary precautions such as rules of thumb) will be applied.

Beginning of the Study:

Participants who meet the study criteria and agree to participate in the study will be randomly assigned to the control group or intervention group.

1. Control group protocol; participants randomized to the control group will not receive any dietary intervention. In this process, how all participants should be asked before starting the study.

   If they are fed, they will be asked to continue in the same way and to maintain their physical activity level.
2. Intervention group protocol; participants randomized to the intervention group will receive a time-restricted feeding intervention for 6 weeks without energy restriction (adlibitum). Meals of the participants will be planned as 8 hours of eating and 16 hours of fasting.

Meal timing will be set as follows:

* First meal at 10:00,
* Last meal at 18:00 in the evening

Participants will be asked not to consume anything other than non-calorie drinks (water, only soda, unsweetened herbal teas, etc.) between 18:00 in the evening and 10:00 in the morning.

ELIGIBILITY:
Inclusion Criteria:

1. 19-65 age range
2. Female
3. BMI: 24.9-29.9 kg/m²
4. Maintaining general activity and exercise habits during the study period
5. Stable body weight (<4 kg weight loss or weight gain) for 6 months prior to the start of the study

Exclusion Criteria:

1. Those with chronic disease (diabetes, hypertension, cardiovascular disease, etc.)
2. Drug users
3. Use of supplements that may affect blood lipid profile and blood sugar (omega-3 etc.)
4. Pregnant women
5. People in the lactation period
6. Menopause
7. Shift workers
8. Those who follow a Time Restricted (16:8) nutrition program before the study
9. Those who have followed any particular diet before the study
10. Those who frequently apply different weight loss diet programs

Ages: 19 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2021-10-24 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
Body Weight | 6 week
  Body Weight
Body Composition | 6 week
  total body fluid
Body Composition | 6 week
  total fat mass
Body Composition | 6 week
  muscle mass
Body Composition | 6 week
  fat free mass
Plasma lipids | 6 week
  Total cholesterol
Plasma lipids | 6 week
  Hdl cholesterol
Plasma lipids | 6 week
  Ldl cholesterol
Plasma lipids | 6 week
  Triglyceride
Blood Pressure | 6 week
  Systolic blood pressure
Blood Pressure | 6 week
  Diastolic blood pressure
Pulse | 6 week
Biochemistry | 6 week
  blood glucose
Biochemistry | 6 week
  fasting insulin

CONTACTS AND LOCATIONS:
Overall Officials: AYŞEN YILDIRIM KIZILDAĞ, PhD, Principal Investigator — Eastern Mediterranean University
Locations (1):
- Eastern Mediterranean University, Famagusta, Cyprus

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 1 year
Access Criteria: No individual participant data will be shared. Results will be published by the investigators in academic journals.